CLINICAL TRIAL: NCT02470195
Title: Anesthesiology Education Implementation by Procedural Simulation Workshop for Difficult Airway Management: a Controlled Interregional French Study
Brief Title: Procedural Simulation for Difficult Airway Training in Anesthesiology Resident Education Program
Acronym: PROSIDIAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, MD, Claude Bernard University
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CLESS PROSIDIAIR 2014
Record Dates: First submitted 2015-05-28; First posted 2015-06-12 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Behaviour
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- workshop (Experimental): workshop of procedural simulation
  Interventions: Behavioral: workshop
- control (No Intervention): no specific workshop of procedural simulation

INTERVENTIONS:
Behavioral: workshop — workshop for procedural simulation for education in difficult airway situation
  Arms: workshop

SUMMARY:
Difficult airway management is a crucial point that may influence outcomes of patient in this critical situation. Education for this topic is of main importance for resident of anesthesiology. Procedural simulation workshop allows participant to use device dedicated to difficult airway management. Investigators included this workshop to a state education program of anesthesiology resident in second year and compared to their homonym in another state where no specific organized workshop is integrated to the education program.

DETAILED DESCRIPTION:
Difficult airway management is a crucial point that may influence outcome of patient in this critical situation. Education for this topic is of main importance for resident of anesthesiology. Procedural simulation workshop allows participant to use device dedicated to difficult airway management. The investigators included this workshop for smal groups of 6-10 anesthesiology resident from Rhône Alpes Auvergne french state. Participants were ask to fill out a questionnaire about their specific knowledge and experience of several devices usable in difficult airway management situation. The workshop was a small briefing as an introduction to the workshop and then small workshop of 20-45 min for specific procedural use of different devices for difficult airway management : Eischmann guide, LMA, supraglottic devices, fiberoptic with spontaneous breathing, cricothyroidotomy, jet ventilation, percutaneous tracheotomy... Investigator will compare at 6 month the incidence of use of the difficult airway devices between resident from rhone alpes auvergne following the workshop and resident from Montpellier that did not follow specific organized workshop.

ELIGIBILITY:
Inclusion Criteria:

* Residents in 2nd year of anesthesiology residency in Rhones alpes auvergne and in Nîmes

Exclusion Criteria:

* Exclusion demand from the participant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
incidence of use of airway devices between groups | 6 month
  modification in the incidence of use of airway devices between workshop and control groups

SECONDARY OUTCOMES:
confidence with airway device | 6 month
  questionnaire of confidence with the usability of the devices. Scale from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: marc Lilot, MD, Principal Investigator — CLESS
Locations (1):
- CLESS, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No
data will be analysed by group, no plan to share data has been programmed

REFERENCES:
- [Derived] Lilot M, Evain JN, Vincent A, Gaillard G, Chassard D, Mattatia L, Ripart J, Denoyel L, Bauer C, Robinson P, Duclos A, Lehot JJ, Rimmele T. [Simulation of difficult airway management for residents: prospective comparative study]. Braz J Anesthesiol. 2019 Jul-Aug;69(4):358-368. doi: 10.1016/j.bjan.2019.02.002. Epub 2019 Jul 29. PMID 31371173